CLINICAL TRIAL: NCT03919617
Title: The Effects of a Glucagon Receptor Antagonist (GRA) on Non-Glucose Metabolic Pathways in Patients With Type 1 Diabetes (Pilot Study)
Brief Title: Metabolic Pathways of GRA in Patients With Type 1 Diabetes
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: REMD Biotherapeutics, Inc. (Industry)
Responsible Party: Principal Investigator, Jeremy Pettus, MD, Assistant Clinical Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UC-MEDJP-02
Record Dates: First submitted 2019-04-15; First posted 2019-04-18 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — volagidemab

STUDY DESIGN:
Intervention Model Description: Single-center, open label, multi-dose study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open-Label REMD-477 (Experimental)
  Interventions: Drug: REMD-477

INTERVENTIONS:
Drug: REMD-477 — 4-Week, open-label, once weekly subcutaneous injection with 70mg REMD-477.

SUMMARY:
A pilot study for individuals with Type 1 Diabetes who are willing to add a GRA (Glucagon Receptor Antagonist) to their current Diabetes treatment regimen. There will be 10 study visits over the course of approximately 8 weeks, with 4 weeks of once weekly, subcutaneous GRA (REMD-477) injection. Testing includes 2 MRI scans, 2 glucose challenges, and 2 insulin withdrawal challenges along with physical assessments and vitals.

DETAILED DESCRIPTION:
This single-center, open label, multi-dose study is designed to elicit pilot data for a larger project. To accomplish the specific aims proposed, a single clinical trial will be conducted in which a maximum of 10 subjects with T1D, who are otherwise healthy, will be treated with REMD-477 for 4 weeks at a dose of 70mg (administered subcutaneously each week) with assessments done pre- and post-therapy. There is no comparator, nor is there any placebo in the study. In addition, there is no randomization, all subjects will receive the same 4 weeks of 70mg, once weekly dose of REMD-477.

There will be 10 study visits as outlined below:

1. Screening - Complete medical history and physical exam, review of current medications, height/weight, vital signs, and fasting laboratory (blood and urine) tests.
2. Visit 1 - Participants that meet screening criteria will be provided deuterated (heavy) water to consume overnight. Participants will ingest heavy water (2H2O) overnight in three equal doses (total 3ml/kg/body water). Participants will also undergo an MRI to evaluate hepatic (liver) fat content as well as total body composition.
3. Visit 2 - Following Visit 1, participants will return to the clinic the next morning in the fasting state (8 hours) and after completing the heavy water consumption. Blood samples will be drawn for baseline amino acid levels as well as samples of serum, plasma, PBMCs, and extracted RNA stored for future metabolomics and genetic testing. Indirect calorimetry (IDC) will be performed to provide baseline resting energy expenditure (REE). Upon completion of IDC, participants will be given a 0.15 u/kg dose of rapid acting insulin and 15 minutes afterwards will ingest a 75g glucose and 25g fructose drink. Participants will then have samples collected over 6 hours to quantify isotope enrichment in plasma water as well as triglyceride isolated from VLDL. Repeat IDC will be performed 2 hours after consumption of the drink.
4. Visit 3 - Insulin withdrawal challenge and injection #1 of REMD-477. Participants will suspend insulin delivery and remove insulin pump. Blood sugars and ketones will be monitored for up to 6 hours.
5. Visit 4 - Injection #2 of REMD-477.
6. Visit 5 - Injection #3 of REMD-477.
7. Visit 6 - Injection #4 of REMD-477.
8. Visit 7 - Provide heavy water and complete MRI scan #2.
9. Visit 8 - Repeat all Visit 2 procedures.
10. Visit 9 - Repeat all Visit 3 procedures.
11. Visit 10 - Safety follow-up visit that includes physical exam, vitals, blood and urine sample collection.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women between the ages of 18 and 65 years old, inclusive, at the time of screening;
2. Females of non-child bearing potential must be ≥ 1 year post-menopausal or documented as being surgically sterile. Females of child bearing potential must agree to use two methods of contraception during the entire study and for an additional 3 months after the end of dosing with the investigational product;
3. Male subjects must be willing to use clinically acceptable method of contraception during the entire study and for an additional 6 months after the end of the treatment period;
4. Diagnosed with Type 1 diabetes based on clinical history or as defined by the current American Diabetes Association (ADA) criteria for > 5 years;
5. Treatment with a stable insulin regimen (< 1u/kg per day) for at least 8 weeks before screening with continuous subcutaneous insulin infusion (CSII) via an insulin pump;
6. HbA1c ≤ 10 % at screening;
7. A minimum weight of 50kg;
8. Able to provide written informed consent approved by an Institutional Review Board (IRB).

Exclusion Criteria:

1. History or evidence of clinically-significant disorder or condition that, in the opinion of the Investigator, would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion;
2. History of pancreatitis, medullary thyroid carcinoma and/or liver disease;
3. Clinically significant diagnosis of anemia;
4. Body Mass Index (BMI) < 18.5 kg/m2 and/or weight less than 50kg;
5. Whole blood donation of 1 pint (500 mL) within 8 weeks prior to Screening. Donations of plasma, packed RBCs, platelets or quantities less than 500 mL are allowed at investigator discretion;
6. Current or recent (within 1 month of screening) use of diabetes medications other than insulin;
7. Women who are pregnant or lactating/breastfeeding;
8. Subjects for whom an MRI is contraindicated;
9. Unable or unwilling to follow the study protocol or who are non-compliant with screening appointments or study visits;
10. Any other condition(s) that might reduce the chance of obtaining study data, or that might cause safety concerns, or that might compromise the ability to give truly informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Change in Beta-hydoxybutyrate (BHB) Level | 4-Weeks
  The change from baseline in peak BHB production as measured by the insulin withdrawal challenge.
Rate of De Novo Lipogenesis (DNL) | 4-Weeks
  Change from baseline in disrupted glucagon signaling as measured by the glucose challenge and deuterated water ingestion.
Rate of Hepatic Steatosis | 4-Weeks
  Changes from baseline in hepatic steatosis as measured by the glucose challenge and deuterated water ingestion.
Rate of Resting Energy Expenditure (REE) | 4-Weeks
  Change from baseline REE as measured by the glucose challenge and deuterated water ingestion.

CONTACTS AND LOCATIONS:
Locations (1):
- UC San Diego Altman Clinical & Translational Research Institute, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No